CLINICAL TRIAL: NCT03459170
Title: A Phase I Study Of Safety, Pharmacokinetics, And Efficacy Of Donor BPX-501 Cells and Rimiducid Infusion For Children With Recurrent Hematologic Malignancies or Minimal Residual Disease After Allogeneic Transplant
Brief Title: Safety/PK Study of Gene Modified Donor T Cell Infusion in Children With Recurrent Hem Malignancies After Allo Transplant
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Bellicum Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BP-I-008
Record Dates: First submitted 2018-02-23; First posted 2018-03-08 (Actual); Last update posted 2022-07-12 (Actual); Status verified 2022-07

CONDITIONS: Hematologic Malignancy
Keywords: leukemia; myelodysplastic syndrome; lymphoma; minimal residual disease; BPX-501; AP1903; rimiducid
MeSH Terms: conditions — Hematologic Neoplasms; Leukemia; Myelodysplastic Syndromes; Lymphoma; Neoplasm, Residual | interventions — AP 1903 reagent

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- BPX-501 T cells and rimiducid (Experimental): All subjects will receive 3 courses of BPX-501 T cell infusions at escalating dose levels (DL). DL1 on Day 0, DL2 on Days 30 and 60. The first dose of BPX-501 T cells will occur ≥30 days after hematopoietic stem cell transplant (HSCT).
  Two doses of AP1903 ( 0.1 mg/kg and 0.4 mg/kg) will be investigated for the treatment of aGvHD after BPX-501 T cell infusion.
  Interventions: Biological: BPX-501 T cells; Drug: rimiducid

INTERVENTIONS:
Biological: BPX-501 T cells — Biological: T cells transduced with CaspaCIDe® safety switch
  Other Names: rivogenlecleucel
Drug: rimiducid — administered to eliminate BPX-501 cells in the event of GVHD
  Other Names: AP1903

SUMMARY:
Phase I, open-label, non-randomized study of safety, pharmacokinetics and efficacy of donor BPX-501 T cell infusion in children with recurrent or minimal residual disease (MRD) hematologic malignancies post-allogeneic transplant. The study will consist of the Main Study and an optional Pharmacokinetics (PK) Sub-Study.

DETAILED DESCRIPTION:
Main Study:

Approximately 16 subjects will participate in the BPX-501 main study. The treatment consists of three courses of BPX-501 T cell infusions at 30 day intervals with 2 escalating dose levels (DL). DL1 on Day 0; DL2 on Days 30 and 60.

Two doses of rimiducid (AP1903) will be investigated for the treatment of aGvHD after BPX-501 T cell infusion. A 0.1mg/kg initial dose of rimiducid which has demonstrated the ability to induce >50% BPX-501 T cell eradication in preclinical animal models will first be administered in the event of uncontrollable aGvHD. If there is no response to this dose within 24hrs + 12hrs a second dose of 0.4 mg/kg (which has been reported to induce T cell eradication of > 90%) will be administered. If there is no measurable GvHD response to the initial dose of 0.1 mg/kg rimiducid in 2 subjects, the starting dose of rimiducid will be 0.4 mg/kg for all subsequent subjects.

Rimiducid (AP1903) Optional PK Sub-Study:

Approximately 12 subjects will be recruited to participate in the optional Rimiducid (AP1903) PK sub-study. Subjects will be assigned to one of two arms and receive either 0.04mg/kg or 0.4mg/kg of Rimiducid (AP1903). Each arm will have a target enrollment of 6 subjects.

* Arm 1: 0.04mg/kg Rimiducid (AP1903), 6 subjects;
* Arm 2: 0.4mg/kg Rimiducid (AP1903), 6 subjects. Rimiducid PK samples and ECG data will be collected at Pre-dose (0 hour), 30 minutes, 2 hours and 8 hours following the initiation of rimiducid (AP1903) infusion.

Efforts shall be made to enroll at least one subject from each age subset into the PK sub-study: infants and toddlers (12 months to 23 months); children (2-11 years); and adolescents (12-18 years).

ELIGIBILITY:
Inclusion Criteria:

* Patients aged < 18
* Clinical diagnosis of one of the following pediatric hematological malignancies:

  * High-risk Acute Leukemia (Acute lymphoblastic leukemia [ALL] or acute myeloid leukemia [AML]) in any CR
  * Acute Leukemia that is minimal residual disease (MRD) positive at > 1copy per 1 x 10,000 reference copies pre-HSCT
  * Myelodysplastic Syndrome (MDS)
  * Hodgkin or Non-Hodgkin lymphomas
  * Other high-risk hematological malignancy in CR eligible for stem cell transplantation per institutional standard
  * Patients with a hematological malignancy who have received a prior allogeneic HSCT
  * Patients with on-treatment relapse of AML within 6 months of initial CR
  * Patients relapsing within 6 months of initial diagnosis of hematological malignancy.
* Planned or previous treatment of hematological malignancy with one of the following:

  * Matched related HSCT
  * Mismatched related HSCT
* For patients who have received a transplant, occurrence of one of the following > 30 days post-HSCT:

  * Minimal residual disease (MRD) positive at > 1 copy per 1 x 10,000 reference copies post-HSCT
  * Decreasing donor chimerism detected on two bone marrow biopsies or peripheral blood analyses at a > 7-day interval
  * Recurrent disease
* Life expectancy >10 weeks;
* Signed donor and patient/guardian informed consent;
* For mismatched related donor recipients, a minimum genotypic identical match of 5/10 is required, as determined by high resolution typing, at least one allele of each of the following genetic loci must be matched: HLA-A, HLA-B, HLA-C, HLA- DRB1, and HLA-DQB1.
* Performance status: Karnofsky/Lansky score > 70%.
* Adequate organ function as measured by:

  * High-risk Acute Leukemia (Acute lymphoblastic leukemia [ALL] or acute myeloid leukemia [AML]) in any CR
  * High-risk Acute Leukemia (Acute lymphoblastic leukemia [ALL] or acute myeloid leukemia [AML]) in any CR
  * Hepatic: direct bilirubin ≤ 3x ULN, or AST/ALT ≤ 5x ULN.
  * Bone marrow;
* > 25% donor T cell chimerism
* ANC >1 x 10^9/L.

  * Cardiac: LVEF at rest >45%.
  * Pulmonary: FEV 1, FVC, DLCO (diffusion capacity for CO) > 50% predicted (corrected for hemoglobin); for children who are unable to perform pulmonary function tests due to age or developmental ability, there must be no evidence of dyspnea or no need for supplemental oxygen as evidenced by 02 saturation ≥ 92% on room air.
  * Hepatic: direct bilirubin ≤ 3x ULN, or AST/ALT ≤ 5x ULN.
  * Renal: creatinine clearance ≤ 2x of ULN for age

Exclusion Criteria:

≥ Grade II acute GVHD or moderate to severe chronic GVHD due to a previous allograft at the time of screening;

* Active CNS involvement by malignant cells (< 2 months prior to time of consent);
* Current uncontrolled bacterial, viral or fungal infection (currently taking medication with evidence of progression of clinical symptoms or radiologic findings).
* Positive HIV serology or viral RNA;
* Pregnancy (positive serum βHCG test) or breast-feeding female;
* Patients of reproductive age unwilling to use effective forms of birth control or abstinence for a year after BPX-501 T cell infusion.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Estimated)
Dates: Start 2018-02-01 (Actual); Primary Completion 2022-09 (Estimated); Study Completion 2035-09 (Estimated)

PRIMARY OUTCOMES:
BPX-501 Safety | Month 24
  Incidence of treatment emergent adverse events of 2 stratified dose levels of BPX-501 T cell infusions based on patient-donor match in pediatric subjects with hematologic malignancies
Mean plasma concentration | pre-dose, 30 min, 2 hours and 8 hours after start of infusion
  Measure plasma concentrations of rimiducid (AP1903) at two doses (Arm 1: 0.04mg/kg; Arm 2: 0.4mg/kg) in pediatric subjects, during and after a 2-hour infusion

SECONDARY OUTCOMES:
Overall survival | Month 24
  Measure overall survival rates after BPX-501 infusion
Response Rate | Month 24
  Assess response rates after BPX-501 infusion

CONTACTS AND LOCATIONS:
Overall Officials: Bellicum Pharmaceuticals, Study Director — Bellicum Pharmaceuticals, Inc.
Locations (3):
- Italy (3):
  - San Matteo Hospital, Pavia
  - IRCCS Ospedale Pediatrico Bambino Gesù, Rome
  - Ospedale Infantile Regina Margherita, Turin